CLINICAL TRIAL: NCT01562444
Title: A Phase IV, Open-label, Single-center Study to Evaluate Long Term Immunogenicity up to 10 Years After the First Booster Immunization With Tick Borne Encephalitis Vaccine in Adults Who Received 1 of 3 Different Primary Vaccination Schedules
Brief Title: Study to Evaluate Long Term Immunogenicity up to 10 Years After the First Booster Immunization With Tick Borne Encephalitis Vaccine in Adults Who Received 1 of 3 Different Primary Vaccination Schedules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 205335; 2011-003255-19 (EudraCT Number); V48P7E2 (Other: Novartis)
Record Dates: First submitted 2012-03-13; First posted 2012-03-23 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Tick Borne Encephalitis; Virus Diseases
Keywords: Long term immunogenicity study
MeSH Terms: conditions — Encephalitis, Tick-Borne; Virus Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TBE_R Group (Other): Subjects who had previously received the Tick borne encephalitis (TBE) primary vaccination according to rapid (R) schedule i.e., on days 0, 7 (+3) and 21 (+7) in the parent study (V48P7) and who were administered 1 booster dose of Encepur adults either 12-18 months after R schedule completion or in the first extension study, V48P7E1 (NCT00387634), were included in this group. Subjects had blood drawn annually starting from year 6 up to year 10 after booster vaccination (for those subjects boostered before V48P7E1 study start, the blood draw occurred annually starting from >6 years up to >10 years after booster vaccination).
  Interventions: Other: Blood draw
- TBE_C Group (Other): Subjects who had previously received the Tick borne encephalitis (TBE) primary vaccination according to conventional (C) schedule i.e., on days 0, 28 (+10) and 300 (+21) in the parent study (V48P7) and were administered 1 booster dose of Encepur adults in the first extension study, V48P7E1 (NCT00387634), were included in this group. Subjects had blood drawn annually starting from year 6 up to year 10 after booster vaccination.
  Interventions: Other: Blood draw
- TBE_AC Group (Other): Subjects who had previously received the Tick borne encephalitis (TBE) primary vaccination according to accelerated conventional (AC) schedule i.e., on days 0, 14 (+3) and 300 (+21) in the parent study (V48P7) and were administered 1 booster dose of Encepur adults in the first extension study, V48P7E1 (NCT00387634), were included in this group. Subjects had blood drawn annually starting from year 6 up to year 10 after booster vaccination.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Annual blood draw at years 6 (Visit 18), 7 (Visit 19), 8 (Visit 20), 9 (Visit 21) and 10 (Visit 22)

SUMMARY:
The aim of this study is to investigate the immunogenicity response in adults up to 10 years after one booster dose. Data collected from this study will allow for greater information to prescribers who administer TBE vaccine, so that they can appropriately time the administration of booster vaccinations to individuals who received different vaccination schedules and who live in tick borne encephalitis endemic regions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed prior study - V48P7E1.

Exclusion Criteria:

* Subjects whose antibody responses to booster vaccine received in the parent study fell below protective levels, subjects who have been exposed to TBE or flavivirus vaccine, subjects with immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2012-03-08 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hradec Králové, Czechia

REFERENCES:
- [Background] Beran J, Lattanzi M, Xie F, Moraschini L, Galgani I. Second five-year follow-up after a booster vaccination against tick-borne encephalitis following different primary vaccination schedules demonstrates at least 10 years antibody persistence. Vaccine. 2019 Jul 26;37(32):4623-4629. doi: 10.1016/j.vaccine.2017.12.081. Epub 2018 Feb 1. PMID 29397225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who completed V48P7E1 study having received primary vaccination according to rapid (R), conventional (C) or accelerated conventional (AC) schedule were included in the study. Since modified conventional (MC) had not been accepted by health authorities as primary vaccination schedule, this group from V48P7 was not enrolled in this study.
Pre-assignment Details: 206 subjects were enrolled in the study but one subject was not assigned to any group. Therefore, the number of subjects started is 205.
Period: Overall Study
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Started | 48 | 51 | 106
Completed | 43 | 49 | 99
Not Completed | 5 | 2 | 7
Not completed — Did not meet entry criteria | 2 | 0 | 3
Not completed — Did not comply with blood draw schedule | 1 | 0 | 1
Not completed — Unavailable serological results | 0 | 2 | 2
Not completed — Protocol forbidden concomitant vaccine | 1 | 0 | 1
Not completed — Protocol forbidden medication | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group | Total
Number analyzed (Participants) | 48 | 51 | 106 | 205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (15.25) | 41.8 (14.34) | 42.4 (14.35) | 42.3 (14.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 32 | 55 | 111
  Male | 24 | 19 | 51 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 51 | 106 | 205

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers Greater Than or Equal to (≥) 2
Description: Antibody titers were measured by GlaxoSmithKline (GSK) neutralizing antibody (NT) assay.
Time Frame: At Year 6
Population: This analysis was performed on All Screened Set which included all subjects who were screened for participation of this study, including screening failures and withdrawals due to insufficient antibody levels or confirmed exposure to a TBE vaccine.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 95.83 [85.75 to 99.49] | 100.0 [93.02 to 100.0] | 97.17 [91.95 to 99.41]

2. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 93.75 [82.80 to 98.69] | 100.0 [93.02 to 100.0] | 95.28 [89.33 to 98.45]

3. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 89.58 [77.34 to 96.53] | 98.04 [89.55 to 99.95] | 93.40 [86.87 to 97.30]

4. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 89.58 [77.34 to 96.53] | 94.12 [83.76 to 98.77] | 92.45 [85.67 to 96.69]

5. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 89.58 [77.34 to 96.53] | 96.08 [86.54 to 99.52] | 93.40 [86.87 to 97.30]

6. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 95.83 [85.75 to 99.49] | 100.0 [93.02 to 100.0] | 97.17 [91.95 to 99.41]

7. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 93.75 [82.80 to 98.69] | 100.0 [93.02 to 100.0] | 95.28 [89.33 to 98.45]

8. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 89.58 [77.34 to 96.53] | 98.04 [89.55 to 99.95] | 92.45 [85.67 to 96.69]

9. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 89.58 [77.34 to 96.53] | 94.12 [83.76 to 98.77] | 92.45 [85.67 to 96.69]

10. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10
Description: Antibody titers were measured by GSK NT assay.
Time Frame: At Year 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Percentage of subjects | 89.58 [77.34 to 96.53] | 94.12 [83.76 to 98.77] | 93.40 [86.87 to 97.30]

11. Primary Outcome: Evaluation of Geometric Mean Antibody Titers (GMTs)
Description: GMTs by visit were tabulated for each vaccine schedule. Baselines pre booster and post booster vaccination titers were used as denominators to calculate Geometric Mean Ratios (GMRs). Pre booster vaccination titer: GMT at Day 0 of V48P7E1 prior to booster vaccine administration (excluding subjects who received the booster before V48P7E1 study start). Post booster vaccination titer: GMT at Day 21 of V48P7E1 (for subjects who received booster in V48P7E1); Day 0 for subjects who received booster before V48P7E1 study start.
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 51 | 104
  Baseline GMT pre booster | 76 [28 to 208] | 228 [149 to 348] | 228 [170 to 307]
  Baseline GMT post booster: number analyzed (Participants) | 48 | 51 | 105
  Baseline GMT post booster | 467 [325 to 670] | 1135 [799 to 1611] | 985 [771 to 1257]
  GMT Year 6 | 292 [184 to 463] | 293 [187 to 458] | 221 [162 to 302]

12. Primary Outcome: Evaluation of GMTs
Description: GMTs by visit were tabulated for each vaccine schedule. Baselines pre booster and post booster vaccination titers were used as denominators to calculate GMRs. Pre booster vaccination titer: GMT at Day 0 of V48P7E1 prior to booster vaccine administration (excluding subjects who received the booster before V48P7E1 study start). Post booster vaccination titer: GMT at Day 21 of V48P7E1 (for subjects who received booster in V48P7E1); Day 0 for subjects who received booster before V48P7E1 study start.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 51 | 104
  Baseline GMT pre booster | 76 [28 to 208] | 228 [149 to 348] | 228 [170 to 307]
  Baseline GMT post booster: number analyzed (Participants) | 48 | 51 | 105
  Baseline GMT post booster | 467 [325 to 670] | 1135 [799 to 1611] | 985 [771 to 1257]
  GMT Year 7 | 295 [180 to 484] | 343 [212 to 555] | 254 [182 to 355]

13. Primary Outcome: Evaluation of GMTs
Description: as for outcome 12
Time Frame: At year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 51 | 104
  Baseline GMT pre booster | 76 [28 to 208] | 228 [149 to 348] | 228 [170 to 307]
  Baseline GMT post booster: number analyzed (Participants) | 48 | 51 | 105
  Baseline GMT post booster | 467 [325 to 670] | 1135 [799 to 1611] | 985 [771 to 1257]
  GMT Year 8 | 134 [79 to 227] | 211 [127 to 352] | 155 [109 to 221]

14. Primary Outcome: Evaluation of GMTs
Description: as for outcome 12
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 51 | 104
  Baseline GMT pre booster | 76 [28 to 208] | 228 [149 to 348] | 228 [170 to 307]
  Baseline GMT post booster: number analyzed (Participants) | 48 | 51 | 105
  Baseline GMT post booster | 467 [325 to 670] | 1135 [799 to 1611] | 985 [771 to 1257]
  GMT Year 9 | 211 [119 to 375] | 214 [122 to 374] | 194 [131 to 285]

15. Primary Outcome: Evaluation of GMTs
Description: as for outcome 12
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 106
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 51 | 104
  Baseline GMT pre booster | 76 [28 to 208] | 228 [149 to 348] | 228 [170 to 307]
  Baseline GMT post booster: number analyzed (Participants) | 48 | 51 | 105
  Baseline GMT post booster | 467 [325 to 670] | 1135 [799 to 1611] | 985 [771 to 1257]
  GMT Year 10 | 166 [94 to 295] | 245 [140 to 428] | 180 [122 to 265]

16. Primary Outcome: Geometric Mean Ratios (GMRs) Calculated to Pre Booster Baselines
Description: GMR values were tabulated by vaccine schedule using pre booster vaccination titers as baseline. Pre booster vaccination titer: GMT at Day 0 of V48P7E1 prior to booster vaccine administration (excluding subjects who received the booster before V48P7E1 study start).
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 51 | 104
Ratios | 6.73 [3.23 to 14.02] | 1.28 [0.94 to 1.75] | 0.99 [0.8 to 1.23]

17. Primary Outcome: GMRs Calculated to Pre Booster Baselines
Description: as for outcome 16
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 51 | 104
Ratios | 3.85 [1.48 to 10] | 1.51 [1.01 to 2.25] | 1.13 [0.85 to 1.5]

18. Primary Outcome: GMRs Calculated to Pre Booster Baselines
Description: as for outcome 16
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 51 | 104
Ratios | 0.67 [0.23 to 1.91] | 0.93 [0.6 to 1.44] | 0.69 [0.51 to 0.95]

19. Primary Outcome: GMRs Calculated to Pre Booster Baselines
Description: as for outcome 16
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 51 | 104
Ratios | 1.08 [0.33 to 3.53] | 0.94 [0.57 to 1.54] | 0.85 [0.6 to 1.21]

20. Primary Outcome: GMRs Calculated to Pre Booster Baselines
Description: as for outcome 16
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 51 | 104
Ratios | 0.76 [0.26 to 2.24] | 1.08 [0.68 to 1.69] | 0.8 [0.59 to 1.1]

21. Primary Outcome: GMRs Calculated to Post Booster Baselines
Description: GMR values were tabulated by vaccine schedule using post booster vaccination titers as baseline. Post booster vaccination titer: GMT at Day 21 of V48P7E1 (for subjects who received booster in V48P7E1); Day 0 for subjects who received booster before V48P7E1 study start.
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 105
Ratios | 0.63 [0.46 to 0.86] | 0.26 [0.19 to 0.35] | 0.22 [0.18 to 0.28]

22. Primary Outcome: GMRs Calculated to Post Booster Baselines
Description: as for outcome 21
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 105
Ratios | 0.63 [0.41 to 0.96] | 0.3 [0.2 to 0.46] | 0.25 [0.19 to 0.34]

23. Primary Outcome: GMRs Calculated to Post Booster Baselines
Description: as for outcome 21
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 105
Ratios | 0.29 [0.18 to 0.47] | 0.19 [0.12 to 0.3] | 0.16 [0.11 to 0.22]

24. Primary Outcome: GMRs Calculated to Post Booster Baselines
Description: as for outcome 21
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 105
Ratios | 0.45 [0.27 to 0.77] | 0.19 [0.11 to 0.32] | 0.2 [0.14 to 0.28]

25. Primary Outcome: GMRs Calculated to Post Booster Baselines
Description: as for outcome 21
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 48 | 51 | 105
Ratios | 0.36 [0.21 to 0.6] | 0.22 [0.13 to 0.36] | 0.18 [0.13 to 0.26]

26. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 2 | 94.29 [80.84 to 99.30] | 100.0 [90.97 to 100.0] | 96.30 [89.56 to 99.23]
  ≥ 50 years: Antibody Titers ≥ 2: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 2 | 100.0 [75.29 to 100.0] | 100.0 [73.54 to 100.0] | 100.0 [86.28 to 100.0]
  ≥ 60 years: Antibody Titers ≥ 2: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 2 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

27. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 2 | 91.43 [76.94 to 98.20] | 100.0 [90.97 to 100.0] | 93.83 [86.18 to 97.97]
  ≥ 50 years: Antibody Titers ≥ 2: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 2 | 100.0 [75.29 to 100.0] | 100.0 [73.54 to 100.0] | 100.0 [86.28 to 100.0]
  ≥ 60 years: Antibody Titers ≥ 2: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 2 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

28. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 2 | 88.57 [73.26 to 96.80] | 97.44 [86.52 to 99.94] | 92.59 [84.57 to 97.23]
  ≥ 50 years: Antibody Titers ≥ 2: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 2 | 92.31 [63.97 to 99.81] | 100.0 [73.54 to 100.0] | 96.00 [79.65 to 99.90]
  ≥ 60 years: Antibody Titers ≥ 2: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 2 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

29. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 2 | 88.57 [73.26 to 96.80] | 92.31 [79.13 to 98.38] | 91.36 [83.00 to 96.45]
  ≥ 50 years: Antibody Titers ≥ 2: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 2 | 92.31 [63.97 to 99.81] | 100.0 [73.54 to 100.0] | 96.00 [79.65 to 99.90]
  ≥ 60 years: Antibody Titers ≥ 2: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 2 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

30. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 2 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 2 | 88.57 [73.26 to 96.80] | 94.87 [82.68 to 99.37] | 92.59 [84.57 to 97.23]
  ≥ 50 years: Antibody Titers ≥ 2: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 2 | 92.31 [63.97 to 99.81] | 100.0 [73.54 to 100.0] | 96.00 [79.65 to 99.90]
  ≥ 60 years: Antibody Titers ≥ 2: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 2 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

31. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 10 | 94.29 [80.84 to 99.30] | 100.0 [90.97 to 100.0] | 96.30 [89.56 to 99.23]
  ≥ 50 years: Antibody Titers ≥ 10: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 10 | 100.0 [75.29 to 100.0] | 100.0 [73.54 to 100.0] | 100.0 [86.28 to 100.0]
  ≥ 60 years: Antibody Titers ≥ 10: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 10 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

32. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Number of subjects
  15-49 years: Antibody Titers ≥ 10 | 91.43 [76.94 to 98.20] | 100.0 [90.97 to 100.0] | 93.83 [86.18 to 97.97]
  ≥ 50 years: Antibody Titers ≥ 10: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 10 | 100.0 [75.29 to 100.0] | 100.0 [73.54 to 100.0] | 100.0 [86.28 to 100.0]
  ≥ 60 years: Antibody Titers ≥ 10: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 10 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

33. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 10 | 88.57 [73.26 to 96.80] | 97.44 [86.52 to 99.94] | 91.36 [83.00 to 96.45]
  ≥ 50 years: Antibody Titers ≥ 10: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 10 | 92.31 [63.97 to 99.81] | 100.0 [73.54 to 100.0] | 96.00 [79.65 to 99.90]
  ≥ 60 years: Antibody Titers ≥ 10: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 10 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

34. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 9
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 10 | 88.57 [73.26 to 96.80] | 92.31 [79.13 to 98.38] | 91.36 [83.00 to 96.45]
  ≥ 50 years: Antibody Titers ≥ 10: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 10 | 92.31 [63.97 to 99.81] | 100.0 [73.54 to 100.0] | 96.00 [79.65 to 99.90]
  ≥ 60 years: Antibody Titers ≥ 10: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 10 | 100.0 [39.76 to 100.0] | 100.0 [29.24 to 100.0] | 100.0 [59.04 to 100.0]

35. Primary Outcome: Percentage of Subjects With Detectable TBE Antibody Titers ≥ 10 by Age Groups
Description: Age groups defined based on age at entry to V48P7E1 study: 15 to 49 years, ≥ 50 years, and ≥ 60 years.
Time Frame: At Year 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Percentage of subjects
  15-49 years: Antibody Titers ≥ 10 | 88.57 [73.26 to 96.80] | 94.87 [82.68 to 99.37] | 92.59 [84.57 to 97.23]
  ≥ 50 years: Antibody Titers ≥ 10: number analyzed (Participants) | 13 | 12 | 25
  ≥ 50 years: Antibody Titers ≥ 10 | 92.31 [63.97 to 99.81] | 91.67 [61.52 to 99.79] | 96.00 [79.65 to 99.90]
  ≥ 60 years: Antibody Titers ≥ 10: number analyzed (Participants) | 4 | 3 | 7
  ≥ 60 years: Antibody Titers ≥ 10 | 100.0 [39.76 to 100.0] | 66.67 [9.43 to 99.16] | 100.0 [59.04 to 100.0]

36. Primary Outcome: Evaluation of GMTs in the Age Group of 15-49 Years
Description: as for outcome 12
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 39 | 79
  Baseline GMT pre booster | 76 [27 to 215] | 253 [153 to 417] | 263 [185 to 375]
  Baseline GMT post booster: number analyzed (Participants) | 35 | 39 | 80
  Baseline GMT post booster | 638 [413 to 984] | 1299 [861 to 1959] | 1008 [757 to 1343]
  GMT Year 6 | 332 [186 to 593] | 341 [197 to 590] | 235 [160 to 344]

37. Primary Outcome: Evaluation of GMTs in the Age Group of 15-49 Years
Description: as for outcome 12
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 39 | 79
  Baseline GMT pre booster | 76 [27 to 215] | 253 [153 to 417] | 263 [185 to 375]
  Baseline GMT post booster: number analyzed (Participants) | 35 | 39 | 80
  Baseline GMT post booster | 638 [413 to 984] | 1299 [861 to 1959] | 1008 [757 to 1343]
  GMT Year 7 | 304 [164 to 564] | 384 [214 to 691] | 250 [166 to 375]

38. Primary Outcome: Evaluation of GMTs in the Age Group of 15-49 Years
Description: as for outcome 12
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 39 | 79
  Baseline GMT pre booster | 76 [27 to 215] | 253 [153 to 417] | 263 [185 to 375]
  Baseline GMT post booster: number analyzed (Participants) | 35 | 39 | 80
  Baseline GMT post booster | 638 [413 to 984] | 1299 [861 to 1959] | 1008 [757 to 1343]
  GMT Year 8 | 151 [80 to 287] | 219 [119 to 402] | 160 [105 to 243]

39. Primary Outcome: Evaluation of GMTs in the Age Group of 15-49 Years
Description: as for outcome 12
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 39 | 79
  Baseline GMT pre booster | 76 [27 to 215] | 253 [153 to 417] | 263 [185 to 375]
  Baseline GMT post booster: number analyzed (Participants) | 35 | 39 | 80
  Baseline GMT post booster | 638 [413 to 984] | 1299 [861 to 1959] | 1008 [757 to 1343]
  GMT Year 9 | 218 [107 to 443] | 211 [108 to 413] | 191 [120 to 305]

40. Primary Outcome: Evaluation of GMTs in the Age Group of 15-49 Years
Description: as for outcome 12
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 81
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 9 | 39 | 79
  Baseline GMT pre booster | 76 [27 to 215] | 253 [153 to 417] | 263 [185 to 375]
  Baseline GMT post booster: number analyzed (Participants) | 35 | 39 | 80
  Baseline GMT post booster | 638 [413 to 984] | 1299 [861 to 1959] | 1008 [757 to 1343]
  GMT Year 10 | 188 [92 to 382] | 266 [136 to 520] | 200 [126 to 319]

41. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 50 Years
Description: as for outcome 12
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 12 | 25
  Baseline GMT pre booster |  | 163 [77 to 348] | 145 [86 to 244]
  Baseline GMT post booster | 201 [111 to 364] | 733 [395 to 1361] | 914 [595 to 1403]
  GMT Year 6 | 207 [107 to 401] | 178 [89 to 355] | 183 [114 to 295]

42. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 50 Years
Description: as for outcome 12
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 12 | 25
  Baseline GMT pre booster |  | 163 [77 to 348] | 145 [86 to 244]
  Baseline GMT post booster | 201 [111 to 364] | 733 [395 to 1361] | 914 [595 to 1403]
  GMT Year 7 | 272 [126 to 588] | 237 [107 to 528] | 270 [155 to 470]

43. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 50 Years
Description: as for outcome 12
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 12 | 25
  Baseline GMT pre booster |  | 163 [77 to 348] | 145 [86 to 244]
  Baseline GMT post booster | 201 [111 to 364] | 733 [395 to 1361] | 914 [595 to 1403]
  GMT Year 8 | 98 [39 to 245] | 189 [73 to 492] | 142 [73 to 275]

44. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 50 Years
Description: as for outcome 12
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 12 | 25
  Baseline GMT pre booster |  | 163 [77 to 348] | 145 [86 to 244]
  Baseline GMT post booster | 201 [111 to 364] | 733 [395 to 1361] | 914 [595 to 1403]
  GMT Year 9 | 193 [74 to 505] | 224 [82 to 609] | 202 [101 to 403]

45. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 50 Years
Description: as for outcome 12
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 12 | 25
  Baseline GMT pre booster |  | 163 [77 to 348] | 145 [86 to 244]
  Baseline GMT post booster | 201 [111 to 364] | 733 [395 to 1361] | 914 [595 to 1403]
  GMT Year 10 | 119 [47 to 302] | 189 [72 to 496] | 129 [66 to 251]

46. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 60 Years
Description: as for outcome 12
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 3 | 7
  Baseline GMT pre booster |  | 64 [13 to 316] | 69 [24 to 197]
  Baseline GMT post booster | 173 [71 to 425] | 573 [203 to 1616] | 498 [253 to 982]
  GMT Year 6 | 189 [52 to 688] | 96 [22 to 427] | 76 [29 to 202]

47. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 60 Years
Description: as for outcome 12
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 3 | 7
  Baseline GMT pre booster |  | 64 [31 to 316] | 69 [24 to 197]
  Baseline GMT post booster | 173 [71 to 425] | 573 [203 to 1616] | 498 [253 to 982]
  GMT Year 7 | 133 [26 to 677] | 120 [18 to 789] | 105 [31 to 360]

48. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 60 Years
Description: as for outcome 12
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 3 | 7
  Baseline GMT pre booster |  | 64 [13 to 316] | 69 [24 to 197]
  Baseline GMT post booster | 173 [71 to 425] | 573 [203 to 1616] | 498 [253 to 982]
  GMT Year 8 | 128 [26 to 620] | 81 [13 to 504] | 71 [21 to 234]

49. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 60 Years
Description: as for outcome 12
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 3 | 7
  Baseline GMT pre booster |  | 64 [13 to 316] | 69 [24 to 197]
  Baseline GMT post booster | 173 [71 to 425] | 573 [203 to 1616] | 498 [253 to 982]
  GMT Year 9 | 224 [52 to 965] | 67 [12 to 362] | 128 [42 to 385]

50. Primary Outcome: Evaluation of GMTs in the Age Group of ≥ 60 Years
Description: as for outcome 12
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Titers
  Baseline GMT pre booster: number analyzed (Participants) | 0 | 3 | 7
  Baseline GMT pre booster |  | 64 [13 to 316] | 69 [24 to 197]
  Baseline GMT post booster | 173 [71 to 425] | 573 [203 to 1616] | 498 [253 to 982]
  GMT Year 10 | 181 [35 to 928] | 57 [9 to 377] | 72 [21 to 248]

51. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 16
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 39 | 79
Ratios | 6.73 [3.02 to 15.01] | 1.35 [0.92 to 1.98] | 0.92 [0.7 to 1.2]

52. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 16
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 39 | 79
Ratios | 3.85 [1.34 to 11.04] | 1.52 [0.92 to 2.52] | 0.96 [0.68 to 1.38]

53. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 16
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 39 | 79
Ratios | 0.67 [0.22 to 2.08] | 0.87 [0.5 to 1.49] | 0.62 [0.42 to 0.91]

54. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 16
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 39 | 79
Ratios | 1.08 [0.3 to 3.88] | 0.84 [0.45 to 1.54] | 0.73 [0.47 to 1.12]

55. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 16
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 9 | 39 | 79
Ratios | 0.76 [0.24 to 2.48] | 1.05 [0.6 to 1.85] | 0.78 [0.52 to 1.16]

56. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 16
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 12 | 25
Ratios |  | 1.09 [0.75 to 1.59] | 1.27 [0.98 to 1.64]

57. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 16
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 12 | 25
Ratios |  | 1.45 [1.01 to 2.1] | 1.87 [1.45 to 2.41]

58. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 16
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 12 | 25
Ratios |  | 1.16 [0.62 to 2.17] | 0.98 [0.63 to 1.52]

59. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 16
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 12 | 25
Ratios |  | 1.37 [0.71 to 2.65] | 1.39 [0.88 to 2.21]

60. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 16
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 12 | 25
Ratios |  | 1.16 [0.63 to 2.12] | 0.89 [0.58 to 1.35]

61. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 16
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 3 | 7
Ratios |  | 1.5 [0.76 to 2.97] | 1.1 [0.7 to 1.72]

62. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 16
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 3 | 7
Ratios |  | 1.88 [0.97 to 3.64] | 1.52 [0.99 to 2.35]

63. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 16
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 3 | 7
Ratios |  | 1.27 [0.44 to 3.66] | 1.03 [0.51 to 2.05]

64. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 16
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 3 | 7
Ratios |  | 1.05 [0.37 to 2.94] | 1.85 [0.94 to 3.64]

65. Primary Outcome: GMRs Calculated to Pre Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 16
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 0 | 3 | 7
Ratios |  | 0.89 [0.39 to 2.06] | 1.04 [0.6 to 1.81]

66. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 21
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 80
Ratios | 0.52 [0.35 to 0.78] | 0.26 [0.18 to 0.38] | 0.23 [0.18 to 0.3]

67. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 21
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 80
Ratios | 0.48 [0.28 to 0.81] | 0.3 [0.18 to 0.49] | 0.24 [0.17 to 0.35]

68. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 21
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 80
Ratios | 0.24 [0.13 to 0.43] | 0.17 [0.1 to 0.3] | 0.16 [0.11 to 0.23]

69. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 21
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 80
Ratios | 0.34 [0.18 to 0.66] | 0.16 [0.09 to 0.3] | 0.19 [0.12 to 0.3]

70. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of 15-49 Years
Description: as for outcome 21
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 35 | 39 | 80
Ratios | 0.29 [0.15 to 0.56] | 0.2 [0.11 to 0.38] | 0.2 [0.13 to 0.3]

71. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 21
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Ratios | 1.03 [0.7 to 1.52] | 0.24 [0.16 to 0.37] | 0.2 [0.15 to 0.27]

72. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 21
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Ratios | 1.36 [0.79 to 2.33] | 0.32 [0.18 to 0.57] | 0.3 [0.2 to 0.44]

73. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 21
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Ratios | 0.49 [0.23 to 1.04] | 0.26 [0.12 to 0.57] | 0.16 [0.09 to 0.27]

74. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 21
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Ratios | 0.96 [0.44 to 2.08] | 0.31 [0.14 to 0.68] | 0.22 [0.13 to 0.39]

75. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 50 Years
Description: as for outcome 21
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 13 | 12 | 25
Ratios | 0.59 [0.28 to 1.24] | 0.26 [0.12 to 0.55] | 0.14 [0.08 to 0.24]

76. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 21
Time Frame: At Year 6
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Ratios | 1.09 [0.47 to 2.55] | 0.17 [0.06 to 0.45] | 0.15 [0.08 to 0.29]

77. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 21
Time Frame: At Year 7
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Ratios | 0.77 [0.21 to 2.86] | 0.21 [0.05 to 0.96] | 0.21 [0.08 to 0.57]

78. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 21
Time Frame: At Year 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Ratios | 0.74 [0.2 to 2.72] | 0.14 [0.03 to 0.64] | 0.14 [0.05 to 0.38]

79. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 21
Time Frame: At Year 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Ratios | 1.29 [0.43 to 3.84] | 0.12 [0.03 to 0.41] | 0.26 [0.11 to 0.58]

80. Primary Outcome: GMRs Calculated to Post Booster Baselines in the Age Group of ≥ 60 Years
Description: as for outcome 21
Time Frame: At Year 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
Number analyzed (Participants) | 4 | 3 | 7
Ratios | 1.05 [0.31 to 3.49] | 0.1 [0.02 to 0.4] | 0.14 [0.06 to 0.36]

ADVERSE EVENTS:
Description: The study was intended to evaluate the persistence of antibody response up to 10 years after booster vaccine administration. Safety profile of the vaccine was not evaluated as per study protocol. Hence, there are no safety results as per planned analysis.
Arm/Group | TBE_R Group | TBE_C Group | TBE_AC Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.